CLINICAL TRIAL: NCT01561248
Title: Repetitive Intestinal Lavage Using Polyethylene Glycol Solution in Patients With EHEC O104:H4 Infection During the German 2011 Outbreak for Prevention of Severe Thrombocytopenia With Subsequently Following Therapeutic Plasmapheresis
Brief Title: Study of Repetitive Intestinal Lavage in Patients With EHEC Associated Hemorrhagic Colitis
Acronym: EHEC-PEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EHEC-2011-PEG
Record Dates: First submitted 2012-01-23; First posted 2012-03-22 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Hemolytic Uremic Syndrome; Hemorrhagic Colitis; Intestinal Infectious Disease; Intestinal Infection Due to E. Coli
Keywords: EHEC; O104:H4; German; outbreak; polyethylene glycol; Bowel lavage
MeSH Terms: conditions — Hemolytic-Uremic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SOC-treatment (No Intervention): Patients with EHEC associated bloody diarrhoea (n=12) receiving standard of care treatment, consisting of intravenous fluids (2-3 liters/daily), analgetics, including paracetamol and metamizol and metoclopramid, if required.
- PEG-Solution, daily bowel lavage (Experimental): Patients with EHEC associated bloody diarrhoea (n=21)receiving SOC-treatment, consisting of i.v. fluids (2-3 liter/day), analgetics ( paracetamol and metamizol) or metoclopramid and orally administered polyethylene glycol-solution daily during the clinical course.
  Interventions: Drug: polyethylene glycol solution for daily bowel lavage.

INTERVENTIONS:
Drug: polyethylene glycol solution for daily bowel lavage. — At admission,patients with severe EHEC infection received two liters of orally administered electrolytes- balanced polyethylene glycol solution for bowel lavage. Treatment was continued with one liter of polyethylene glycol solution daily for repetitive intestinal lavage during the clinical course.
  Other Names: Klean-Prep(Norgine GmBH, Marburg, Germany).
  Arms: PEG-Solution, daily bowel lavage

SUMMARY:
The investigators examined the outcome of patients with severe Enterohaemorrhagic E. Coli (EHEC) O104:H4 infection suffering from bloody diarrhoea that were at risk to develop hemolytic uremic syndrome and underwent repetitive whole bowl lavage during hospitalization.

DETAILED DESCRIPTION:
During the 2011 German EHEC O104:H4 outbreak, centered in the area of Hamburg, 33 patients with EHEC associated hemorrhagic colitis were admitted to the first Department of Medicine of the Hamburg University medical centre.

The first 12 patients were treated symptomatically and received intravenous rehydration up to three liters daily.

Prompted by a good clinical response after whole bowel irrigation with polyethylene glycol-solution (PEG)in patient 13 all subsequent admitted patients (n=21) were treated with PEG-solution ( 2 liters on admission followed by one liter per day during the clinical course).

During the hospital course blood work was obtained every day and patients were examined for clinical symptoms.

Thrombocytopenia below 100.000/microliter was defined as a threshold for initiating therapeutic plasmapheresis to prevent the onset of hemolytic syndrome on an early stage.

ELIGIBILITY:
Inclusion Criteria:

* Proven EHEC O104:H4-infection

Presence of bloody diarrhoea + at least one of the following serological criteria:

* platelet count below 150x10³/ μl but greater than 100x10³/ μl, serum creatine above normal level for age (> 1.1 -1.3 mg/dl), Lactate dehydrogenase (LDH) > 300 IU/l, leukocytosis ( > 12x10³/ μl ) and elevated CRP (> 5mg/l), hemoglobin < 13.8 g/dL for male patients or < 12.1 g/dL for female patients, respectively or decrease in haptoglobin

Exclusion Criteria:

* Bloody diarrhoea due to others reasons than EHEC O104:H4 infection
* Thrombocytopenia < 100x10³/ μl.
* HUS, defined as platelet count below 100x10³/ μl, anaemia or decrease in haptoglobin and serum creatine above normal level for age

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Thrombocytopenia (Defined as platlet count below 100.000/microliter) | Patients will be followed for the duration of hospital stay, an expected average of two weeks
  Following admission, blood samples were taken every day during the hospital course. When a platelet count below 100.000/microliter was measured, patients were subsequently transfered to the department of nephrology for therapeutic plasmapheresis.
  As thrombocytopenia is the first abnormal laboratory finding in EHEC infected patients developing HUS, therapeutic plasmapheresis was initiated to prevent onset of mature HUS when thrombocytopenia (defined as mentioned above )was measured.

SECONDARY OUTCOMES:
Duration of hospitalisation | Patients will be followed for the duration of hospital stay, an expected average of two weeks
  Secondary outcome in this study was the duration of hospitalisation in the two groups. Duration of hospitalisation was assessed by reviewing the case notes.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Lüth, M.D., Study Director — Department of Medicine, University Medical Centre Hamburg-Eppendorf, Hamburg; Thorben Fründt, M.D., Principal Investigator — Department of Medicine, University Medical Centre Hamburg-Eppendorf, Hamburg
Locations (1):
- 1Department of Medicine, University Medical Centre Hamburg-Eppendorf, Hamburg, Hamburg, Hamburg, Germany